CLINICAL TRIAL: NCT05529160
Title: A Prospective, 1-Arm, Open Label, Non-Randomized Study of the FERTI-LILY Conception Cup Device to Assess Label Comprehension, Device Usability and Safety in Women
Brief Title: FERTI-LILY Safety Study
Status: Completed | Type: Observational
Sponsor: Rosesta Medical BV (Industry)
Responsible Party: Sponsor
Other Study IDs: FCC-001
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2022-09

CONDITIONS: Natural Conception; Label Comprehension; Device Usability; Safety Issues

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Population: Up to 20 subjects will be recruited from the patient population at the Principal Investigator's clinic. Subject recruitment will end once 15 evaluable subjects have completed the study.
  Interventions: Device: FERTI LILY Conception Cup

INTERVENTIONS:
Device: FERTI LILY Conception Cup — The FERTI-LILY Conception Cup is indicated for over-the-counter (OTC) home use by couples trying to conceive. The FERTI·LILY device OTC contains a cervical cap attached to a stem. The FERTI-LILY Conception Cup is intended to push semen towards the cervix as an aid in conception. It is designed to be inserted vaginally after intercourse and left in place for 20-60 minutes. The device is recommended to be used during the ovulatory phase of the menstrual cycle. It is not to be left in place for longer than six hours. The device may be re-used up to 18 times or over 6 cycles.

SUMMARY:
The study is a prospective, 1-arm, open label, nonrandomized, single center study designed to evaluate label comprehension, device usability and safety of the FERTI·LILY Conception Cup. The primary safety endpoint will be an assessment of reported adverse events.

Subjects will be screened -10 (±3) days prior to the baseline visit. At baseline, 15-20 subjects meeting the inclusion/exclusion criteria will be provided with a FERTI·LILY Conception Cup device and instructions for using the device. Subjects will participate in a label comprehension protocol that includes the physician confirmation that they have adequate comprehension to enroll. If not, a screen failure form is completed.

Subjects will agree to try and use the device within 2 weeks of disposition therefore at baseline a two-week visit is scheduled. In the event they do not use the device within the two-week period the follow up visit can be rescheduled based on the visit window of +14 days. If it is not used within 4 weeks, the PI will have the subject return to the site to authorize another two-week period that will be captured as unscheduled follow up visit. The subject should complete the Device Experience Survey after each device use. The Device Experience Survey will be returned at this time, and adverse events will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female volunteer, age ≥ 18 years.
* Subject is willing and able to provide written informed consent for study participation.
* Subject agrees to use the FCC device as directed.
* Subject agrees to complete all study-related assessments.
* Subject agrees to try to use the cup within two weeks of disposition.
* PI confirms that the subject had the adequate label comprehension to enroll in the study.

Exclusion Criteria:

* Subject has a medical condition or other factor that, in the opinion of the investigator, would contraindicate participation in the study.
* Subject has active bacterial vaginosis infection or vaginismus.
* Subject has an abnormal clinically significant Pap Smear diagnosis.
* Subject has a history of endometriosis.
* Subject has any contraindications with the Instructions for Use.
* Subject has an allergy to silicone.
* Subject is pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject is a female volunteer, age ≥ 18 years.
Study Population: Subjects who meet study eligibility criteria will be recruited from the patient population of the Principle Investigator's clinic.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Safety of Device | 6 weeks
  Occurrence of device-related adverse events.

SECONDARY OUTCOMES:
Label Comprehension Assessment Protocol | 6 weeks
  PI using questions and answers to assess comprehension and confirms subject can specify location and use of cup in vaginal model.
Device Usability | 6 weeks
  After use reported by subject: ease of use, user compliance, overall satisfaction, comfort, size of device.

CONTACTS AND LOCATIONS:
Locations (1):
- Boca Raton Obstetrics and Gynecology, Boca Raton, Florida, United States